CLINICAL TRIAL: NCT03991208
Title: Malarone Pharmacokinetics Under Simulated Physiologic Stressors of Deployment
Acronym: MPUSPSD
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to recruit
Sponsor: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Walter_Reed
Record Dates: First submitted 2019-06-14; First posted 2019-06-19 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Exercise; Pharmacokinetics
Keywords: Pharmacokinetics; Exercise; Malaria Prophylaxis; Bioequivalence; Bioavailability
MeSH Terms: conditions — Motor Activity | interventions — atovaquone, proguanil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Rest (Experimental): Pharmacokinetics of Single Dose Malarone at Rest
  Interventions: Drug: Malarone
- Exercise (Experimental): Pharmacokinetics of Single Dose Malarone under exercise in a heat chamber
  Interventions: Drug: Malarone

INTERVENTIONS:
Drug: Malarone — Malarone

SUMMARY:
A 2x2 randomized crossover of single dose malarone at rest and during moderate intensity exercise under controlled conditions of heat and humidity in healthy adult participants. Statistical analysis of AUC and Cmax will be performed to determine pharmacokinetic changes.

DETAILED DESCRIPTION:
A clinical trial under controlled heat exposure and moderate intensity exercise, determined by VO2max testing and calibration, to determine if physiologic changes during heat exposure and exercise change the pharmacokinetics of malarone to a degree that falls outside the range of that which is considered bioequivalent or 80-125% concentration using AUC and Cmax for rate and extent of exposure. Participants will be randomized to order of rest and exercise components. Single dose malarone will be used during both arms. Single dose malarone pharmacokinetics will give insight into risk of toxicity or risk of under treatment during prophylaxis administration.

ELIGIBILITY:
Inclusion Criteria:

Healthy adult female and male ages 18-44 weighing greater than 40kg with BMI less than 30.

Exclusion Criteria:

17 years old or younger, 45 years old or older, unable to speak and read English, unable to perform exercise tests safely, and/or unable to consent to participate. Unwilling to undergo blood draws. Have known allergy to sunflower butter or are unwilling or unable to consume 2 tbsp or have an allergy to any component of malarone. Also non abstinent females at risk of becoming pregnant or in a heterosexual sexual relationships must be willing to use there chosen and available form of contraception defined as barrier protection, implantable device or hormones, or oral contraceptive pills during time of study up to 2 months after or abstinence unless previously sterile with tubal ligation 1 year or greater prior to screening or hysterectomy.

Those with any of the following conditions will also be excluded from the study: history of any of the following: rhabdomyolysis or heat stroke, heart disease, pulmonary disease, chronic kidney disease, single kidney, chronic hepatitis, diabetes, seizure disorders, multiple sclerosis, COPD, asthma, sickle cell trait or disease, thalassemia, thyroid disease, cancer, chronic infections such as history of HIV, HEP B or HEP C, or rheumatologic disorder; current pregnancy or lactation, systolic blood pressure over 140 mm Hg or diastolic pressure over 90 mm Hg; anemia (hematocrit lower than 36% for women and 38% for men and hemoglobin below 11g/dL for women and 12g/dL for men); diabetes (blood glucose above 110 mg/dL); use of any medications for chronic medical conditions (such as glucose-lowering drugs, prednisone, or beta blockers); or any condition that leads to inability to run safely on a treadmill. Non systemic drugs for skin condition or seasonal allergies will not be a disqualifier. Any volunteers identified during the cardiac risk assessment as above low risk will also be excluded from the study. The ACSM guidelines for exclusion criteria identify low-risk individuals as younger than 45, without history of CVD, and with no more than one risk factor according to the ACSM Risk Stratification Questionnaire for stratification. Risk factors include family history of heart disease, smoking status, hypertension with a blood pressure above 140/90, hypercholesterolemia with cholesterol over 200 mg/dL, fasting glucose over 110 mg/dL, obesity with a percent body fat >25% for men or > 30% for women, and (be consistent throughout including ICD) sedentary lifestyle. The monitoring physician can also exclude a volunteer based on his or her medical opinion given the results of a physical exam and/or EKG results.

Initial screening for history will be performed by phone interview with requested waived consent. Those not able to achieve 80% pass on ICD test in 2 tries or less.

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-24 (Estimated); Primary Completion 2021-05-23 (Estimated); Study Completion 2021-05-23 (Estimated)

PRIMARY OUTCOMES:
AUC | 216 hours
  Area Under the Curve of Atovaquone, Proguanil, Cycloguanil
Cmax | 216 hours
  Cmax of Atovaquone, Proguanil, Cycloguanil

CONTACTS AND LOCATIONS:
Locations (1):
- Uniformed Services University, Bethesda, Maryland, United States